CLINICAL TRIAL: NCT07386587
Title: Response of Methotrexate Alone Versus Methotrexate Combined With Etanercept for Achieving Minimal/Low Disease Activity in Patients of Juvenile Idiopathic Arthritis
Brief Title: Methotrexate Alone vs Methotrexate + Etanercept for Minimal/Low Disease Activity in Juvenile Idiopathic Arthritis
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: University of Child Health Sciences and Children's Hospital, Lahore (Other)
Responsible Party: Principal Investigator, Dr Faisal Haneef, Post Graduate Trainee, University of Child Health Sciences and Children's Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 914/CH-UCHS
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: JIA
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Injections; Etanercept; Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Masking Description: This is an open label study, No masking both the participants and the investigators, including care providers and outcome assessors, are aware of the treatment assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A Includes those patients who fulfills inclusive criteria and given Tablet methotrexate 10-15mg/m2/week orally along with Injection Etanercept 0.8mg/kg/week subcutaneously.
  Interventions: Drug: Injection, Etanercept, 25 Mg (Code May Be Used for Medicare When Drug Administered Under the Direct Supervision of A Physician, Not for Use When Drug is Self Administered)
- Group B (Active Comparator): Group B Includes those patients who fulfills inclusive criteria and given Tablet methotrexate 10-15mg/m2/week orally alone
  Interventions: Drug: Injection, Etanercept, 25 Mg (Code May Be Used for Medicare When Drug Administered Under the Direct Supervision of A Physician, Not for Use When Drug is Self Administered)

INTERVENTIONS:
Drug: Injection, Etanercept, 25 Mg (Code May Be Used for Medicare When Drug Administered Under the Direct Supervision of A Physician, Not for Use When Drug is Self Administered) — Injection Etanercept is biological TNF Inhibitor.

SUMMARY:
This open labelled randomized controlled trial will be carried out at the University of Child Health and the Children's Hospital, Lahore consisting of 6 months . In total 60 patients (30 in each group) fulfilling the inclusion criteria will be selected and enrolled in this study. Patients will be divided into two groups; Group A (Injection Etanercept+ Tab methotrexate) and Group B (Injection Etanercept+ Tab methotrexate).

Data will be collected at baseline, 1,3 and 6 months. Data will be collected and recorded

DETAILED DESCRIPTION:
Juvenile Idiopathic Arthritis (JIA) is the primary form of inflammatory arthritis observed in children. JIA is characterized by inflammation of the synovial tissue, which is present in joints, around tendons. The treatment approach for JIA depends on the specific subtype and severity of the disease. It involves the use of various medications, including non-steroidal anti-inflammatory drugs (NSAIDs), oral and intra-articular corticosteroids, as well as both biologic and nonbiologic disease-modifying anti-rheumatic drugs (DMARDs). This open labelled randomized controlled trial will be carried out at the University of Child Health and the Children's Hospital, Lahore consisting of 6 months after approval. In total 60 patients (30 in each group) fulfilling the inclusion criteria will be selected and enrolled in this study. Patients will be divided into two groups; Group A (Injection Etanercept+ Tab methotrexate) and Group B (Tab methotrexate Monotherapy).

Data will be collected at baseline, 1,3 and 6 months. Data will be collected and recorded on a performa. Data will be analyzed through SPSS version 26. For quantitative variables, mean and standard deviation will be calculated and for qualitative variables frequency and percentages will be calculated. chi-square test will be used to estimate the association between qualitative variables. A p-value<0.05 will be significant. The primary goal of this study is to reduce the duration of active arthritis, improve the quality of life for both patients and their parents, and minimize the risk of irreversible osteoarthritic changes

ELIGIBILITY:
Inclusion Criteria:

Polyarticular JIA patients aged 2-16years Male or female patients Newly diagnosed patients

Exclusion Criteria:

Other type of JIA including systemic-onset JIA, psoriatic arthritis, enthesitis-related arthritis, and oligoarticular arthritis Chronic or acute infection or severe infection episodes that required hospitalization or intravenous administration of antibiotics 30 days prior to study initiation A previous history of malignancy Active tuberculosis or any opportunistic infection, including herpes zoster Hepatitis B Positive patients A history of any chronic disease (except for JIA) that could influence the effectiveness or safety of the investigational medicinal product in investigator's opinion

-

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-27 (Actual); Primary Completion 2026-07-27 (Estimated); Study Completion 2026-07-27 (Estimated)

PRIMARY OUTCOMES:
Achievement of Minimal/Low Disease Activity Level in Polyarticular JIA | 24 weeks
  Proportion of patients achieving minimal/Low disease activity based on JDAS-10 between 0.8 t0 3.9 in Polyarticular Juvenile Idiopathic Arthritis.

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Haneef, Principal Investigator — University of Child Health Sciences Lahore.
Locations (1):
- University of Child Health Sciences Lahore, The Children's hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because of participants consent.